CLINICAL TRIAL: NCT07071480
Title: Noninvasive Therapeutic Hypothermia for Tinnitus
Brief Title: Noninvasive Therapy for Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Restorear Devices LLC (Industry)
Collaborators: University of Miami (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250377; 1R43DC022211-01A1 (NIH)
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Tinnitus; Tinnitus, Subjective
Keywords: tinnitus; ringing; ringing in the ears; subjective tinnitus; constant tinnitus; treatment; symptom reduction; symptom management; tinnitus management; intervention
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Mild Therapeutic Hypothermia (MTH) Arm (Experimental): Subjects will receive hypothermia treatment delivered with ReBound devices, applied in a single 30 minute session in-clinic. Baseline audiometric testing and subjective tinnitus assessment will be measured prior to initiation of the treatment. Testing will be repeated immediately after treatment, and changes will be noted. Subjects in this group will also be sent home with a device to use as needed for a period of 6 months. They will be asked to complete monthly subjective surveys online assessing tinnitus severity and monitoring potential adverse events. MTH Arm will complete both Aims 1 and 2. n=20.
  Interventions: Device: Cold pack-delivered mild therapeutic hypothermia
- Control Arm (Sham Comparator): Subjects will receive a sham wearable headband in a single 30 minute session in-clinic. Baseline audiometric testing and subjective tinnitus assessment will be measured prior to initiation of the treatment. Testing will be repeated immediately after treatment, and changes will be noted. Subjects in this group will also be sent home with a device to use as needed for a period of 6 months. They will be asked to complete monthly subjective surveys online assessing tinnitus severity and monitoring potential adverse events. Control Arm will complete both Aims 1 and 2. n=20.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Cold pack-delivered mild therapeutic hypothermia — Mild therapeutic hypothermia (cooling), delivered non-invasively to the structures of the inner ear (cochlea) for 30 minutes, using headband-style proprietary device, ReBound.
  Arms: Mild Therapeutic Hypothermia (MTH) Arm
Device: Sham device — Sham headband-style device. Participants assigned to use this device will be told they are receiving therapy for 30 minutes. However, no therapy is being provided.
  Arms: Control Arm

SUMMARY:
The goal of this interventional clinical study is to establish mild therapeutic hypothermia, delivered non-invasively to the structures of the inner ear, as a safe and repeatable therapeutic method for symptomatic relief of tinnitus. The study will assess both objective and subjective measures to address two main aims:

1. Ascertain the benefits of mild therapeutic hypothermia for symptomatic relief of chronic tinnitus in participants using the ReBound hypothermia device.
2. Ascertain the benefits of mild therapeutic hypothermia for symptom management in chronic tinnitus participants over six months using the ReBound device.

Participants will wear the ReBound hypothermia device for 30 minutes in a single session. Researchers will compare results from those receiving the therapy to those from a control group (sham therapy). Participants will also use the device in-home for 6 months and monitor their symptoms with online surveys.

DETAILED DESCRIPTION:
Tinnitus is the perception of sound in the absence of an external stimulus commonly described as ringing in the ears. Tinnitus is a highly common condition, with most individuals experiencing it at some point in their lifetime. At least 1 in 10 US adults experience chronic or disabling tinnitus [1] with a significant negative impact on quality of life, often affecting sleep, concentration, mood, and hearing ability. Tinnitus can be intermittent or constant in nature, and intensity can vary or be exacerbated by stress, noise exposure, or other factors. Currently, there is no widely applicable cure for tinnitus, and management typically includes use of sound therapy, mental health counseling, lifestyle modifications, stress management, and distraction techniques, all of which serve to mask symptoms without addressing underlying physiology. Tinnitus is associated with changes in auditory function, with hearing loss being the most associated co-morbidity in patients. However, tinnitus can also be observed in patients with audiometrically normal hearing [2, 3].

Tinnitus can have a significant deleterious effect on a person's quality of life, and there is currently no cure. State-of-the art treatment options suffer limitations and are often ineffective and complex. Most widely used tinnitus treatments focus on reducing awareness of tinnitus/masking symptoms and the impact on emotional state rather than seeking to address the underlying mechanisms of the sound generation [4]. Treatment modalities include sound therapy using environmental sounds and/or hearing aids, psychological interventions including tinnitus retraining therapy and/or cognitive behavioral therapy, somatosensory stimulation including vagus nerve stimulation and osteopathic manipulation, and distraction exercises including guided breathing and development of new hobbies. Other therapies aim to target the generation of tinnitus, including direct and indirect stimulation of the auditory cortex and/or other brain structures through neuromodulation and pharmacologics [5]. Despite the limited success of many of these treatment modalities, none have been shown to be widely applicable to manage tinnitus severity or provide a treatment for tinnitus. Further, systematic reviews have failed to demonstrate a strong evidence base for these approaches [1]. Many treatments and strategies currently in research are costly in terms of both time and resources, reducing sufferers' access or their ability to continue treatment over time. For those who do not find relief from their debilitating symptoms, and for those seeking to address secondary effects of tinnitus, there exists a need for novel treatment aimed at reducing acute tinnitus severity [6].

The investigators propose to show the efficacy of a highly accessible and translatable, non-invasive device utilizing mild therapeutic hypothermia, or MTH, to reduce tinnitus severity in participants with tinnitus. Unlike other approaches, MTH will address the physiological mechanisms of tinnitus and is easily deployable for routine use and symptom management. With support from a prior SBIR Phase I award, the investigators have designed and manufactured the headband-style device, ReBoundTM, to provide therapeutic hypothermia to the inner ear structures. Modifying temperature of the cochlea is known to influence auditory responses [7-12]. The investigators and others have shown that MTH delivered locally or systemically protects hearing function and cochlear structures against noise-induced hearing loss when compared to normothermic animals [13]. The present study builds upon strong preliminary and published results of MTH treatment in the inner ear [14, 15] and two additional new publications [16, 17].

The goal of this interventional clinical study is to establish mild therapeutic hypothermia, delivered non-invasively to the structures of the inner ear, as a safe and repeatable therapeutic method for symptomatic relief of tinnitus. The study will assess both objective and subjective measures to address two main aims:

1. Ascertain the benefits of mild therapeutic hypothermia for symptomatic relief of chronic tinnitus in participants using the ReBound hypothermia device.
2. Ascertain the benefits of mild therapeutic hypothermia for symptom management in chronic tinnitus participants over six months using the ReBound device.

Participants will wear the ReBound hypothermia device for 30 minutes in a single session. Researchers will compare results from those receiving the therapy to those from a control group (sham therapy). Participants will also use the device in-home for 6 months and monitor their symptoms with online surveys.

This research will be highly impactful given the significant adverse effects of tinnitus, an unmet clinical need, on a broad population, and the high translational potential of MTH for reducing tinnitus symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older at the time of signing the consent form
* Fluency in English or Spanish
* Chronic subjective tinnitus for more than 30 days defined as audible at least 75% of waking hours
* At least mild tinnitus, score ≥18 on the Tinnitus Handicap Inventory (THI)

Exclusion Criteria:

* Severe anxiety, score ≥ 15 on the Generalized Anxiety Disorder-7 (GAD-7)
* Tinnitus described as non-auditory or pulsatile in nature
* Catastrophic tinnitus, score ≥78 on the THI
* Tinnitus that is intermittent in nature
* Abnormal tympanometric findings
* Presence of conductive component as characterized by air-bone gaps ≥15 dB at two or more consecutive frequencies
* Otologic pathologies (including, but not limited to): acoustic neuroma/ vestibular schwannoma, chronic ear disease, Meniere's disease, documented fluctuating hearing loss, or ototoxicity
* Temporomandibular joint disorder
* Those who are currently receiving medical, pharmacologic, or therapeutic intervention for tinnitus or other otologic conditions.
* Active hearing aid use
* Dizziness at the time of signing the consent form or at the time of starting the study protocol treatment
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) of Tinnitus Severity | VAS will be given to participants in both Experimental and Sham Arms. For Aim 1, VAS will be administered at baseline, immediately after treatment, and at 24 hours post-treatment. For Aim 2, VAS will be administered monthly for 6 months post-baseline.
  3-item instrument used to assess participant's subjective perception of tinnitus. Includes sliding scales used by participants to score their perceived disease severity. VAS will be used to assess perceived tinnitus severity before baseline treatment and repeated immediately after treatment. The VAS consists of a sliding scale from 0 to 10, with 10 correlating to a greater disease burden/worse symptoms.
Tinnitus Functional Index Adapted (TFI-Adapted) | TFI-Adapted will be given to participants in Aim 1. TFI-Adapted will be administered at baseline and 24 hours post-treatment.
  25-item instrument with eight subscales; (1) Intrusiveness, (2) Sense of control, (3) Cognition, (4) Sleep, (5) Auditory, (6) Relaxation, (7) Quality of life, and (8) Emotional distress. Each subscale can be scored separately, allowing for relevant items to be summed and weighted for analysis. TFI questions will be adapted to ask participants about their tinnitus experience over the past 24 hours.

SECONDARY OUTCOMES:
Pure Tone Audiometry | PTA will be measured in Aim 1 at baseline and immediately after treatment.
  PTA will be measured in Aim 1 for frequencies 250 - 8,000 Hz and high frequencies of > 8,000 Hz.
Distortion Product Otoacoustic Emissions (DPOAE) | DPOAE will be measured in Aim 1 at baseline and immediately after treatment.
  DPOAE will be measured in Aim 1 for 1,500 - 10,000 Hz. DPOAEs will be recorded and analyzed using f2 tone frequencies with a fixed primary ratio (f2/f1) of 1.22, L1 = 65 dB SPL, L2 = 55 dB SPL.
Auditory Brainstem Response (ABR) | ABR will be measured in Aim 1 at baseline and immediately after treatment.
  Test measuring the brain's electrical activity in response to sound to assess hearing and neurological function. ABR will be recorded using 77 dB nHL. At least 2 averaged responses will be performed to ensure replicability.
Tinnitus Pitch & Loudness Matching | Tinnitus pitch and loudness matching will be measured in Aim 1 at baseline and immediately after treatment.
  Psychoacoustic measurements of each participant's tinnitus will be performed to qualify tinnitus pitch.
Tinnitus Functional Index (TFI) | TFI will be given to participants in Aim 2. TFI will be administered monthly for 6 months post-baseline.
  25-item instrument with eight subscales; (1) Intrusiveness, (2) Sense of control, (3) Cognition, (4) Sleep, (5) Auditory, (6) Relaxation, (7) Quality of life, and (8) Emotional distress. Each subscale can be scored separately, allowing for relevant items to be summed and weighted for analysis.

OTHER OUTCOMES:
Tinnitus Handicap Inventory (THI) | The THI will be administered as part of enrollment determination and at 6 months post-baseline.
  25-item instrument used to assess the handicap experienced by the participant due to tinnitus. THI assesses functional, emotional, and catastrophic response reactions to tinnitus on a 4-point scale totaling 100, with degree of handicap increasing with score.
Tinnitus Therapy Use | This instrument will be administered monthly for 6 months post-baseline.
  2-question survey to collect data on the number of times the ReBound device was worn in the past month.
Adverse Event Questionnaire (AEQ) | AEQ will be administered immediately after treatment, 24 hours post-treatment, and monthly for 6 months post-baseline.
  2-question survey to collect data on any adverse event associated with use of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Suhrud M Rajguru, PhD, Principal Investigator — RestorEar Devices
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rincon Sabatino S, Rivero A, Sangaletti R, Dietrich WD, Hoffer ME, King CS, Rajguru SM. Targeted therapeutic hypothermia protects against noise induced hearing loss. Front Neurosci. 2024 Jan 16;17:1296458. doi: 10.3389/fnins.2023.1296458. eCollection 2023. PMID 38292902
- [Background] Rincon Sabatino S, Sangaletti R, Griswold A, Dietrich WD, King CS, Rajguru SM. Transcriptional response to mild therapeutic hypothermia in noise-induced cochlear injury. Front Neurosci. 2024 Jan 17;17:1296475. doi: 10.3389/fnins.2023.1296475. eCollection 2023. PMID 38298897
- [Background] Tamames I, King C, Huang CY, Telischi FF, Hoffer ME, Rajguru SM. Theoretical Evaluation and Experimental Validation of Localized Therapeutic Hypothermia Application to Preserve Residual Hearing After Cochlear Implantation. Ear Hear. 2018 Jul/Aug;39(4):712-719. doi: 10.1097/AUD.0000000000000529. PMID 29240567
- [Background] Tamames I, King C, Bas E, Dietrich WD, Telischi F, Rajguru SM. A cool approach to reducing electrode-induced trauma: Localized therapeutic hypothermia conserves residual hearing in cochlear implantation. Hear Res. 2016 Sep;339:32-9. doi: 10.1016/j.heares.2016.05.015. Epub 2016 May 31. PMID 27260269
- [Background] Henry KR. Hyperthermia exacerbates and hypothermia protects from noise-induced threshold elevation of the cochlear nerve envelope response in the C57BL/6J mouse. Hear Res. 2003 May;179(1-2):88-96. doi: 10.1016/s0378-5955(03)00097-2. PMID 12742241
- [Background] Watanabe F, Koga K, Hakuba N, Gyo K. Hypothermia prevents hearing loss and progressive hair cell loss after transient cochlear ischemia in gerbils. Neuroscience. 2001;102(3):639-45. doi: 10.1016/s0306-4522(00)00510-8. PMID 11226700
- [Background] Henry KR, Chole RA. Hypothermia protects the cochlea from noise damage. Hear Res. 1984 Dec;16(3):225-30. doi: 10.1016/0378-5955(84)90111-4. PMID 6401081
- [Background] Ohlemiller KK, Siegel JH. Cochlear basal and apical differences reflected in the effects of cooling on responses of single auditory nerve fibers. Hear Res. 1994 Nov;80(2):174-90. doi: 10.1016/0378-5955(94)90109-0. PMID 7896576
- [Background] Ohlemiller KK, Siegel JH. The effects of moderate cooling on gross cochlear potentials in the gerbil: basal and apical differences. Hear Res. 1992 Nov;63(1-2):79-89. doi: 10.1016/0378-5955(92)90076-y. PMID 1464578
- [Background] Liberman MC, Dodds LW. Single-neuron labeling and chronic cochlear pathology. II. Stereocilia damage and alterations of spontaneous discharge rates. Hear Res. 1984 Oct;16(1):43-53. doi: 10.1016/0378-5955(84)90024-8. PMID 6511672
- [Background] Brown MC, Smith DI, Nuttall AL. The temperature dependency of neural and hair cell responses evoked by high frequencies. J Acoust Soc Am. 1983 May;73(5):1662-70. doi: 10.1121/1.389387. PMID 6863743
- [Background] Kleinjung T, Langguth B. Avenue for Future Tinnitus Treatments. Otolaryngol Clin North Am. 2020 Aug;53(4):667-683. doi: 10.1016/j.otc.2020.03.013. Epub 2020 May 4. PMID 32381341
- [Background] Eggermont JJ, Roberts LE. The neuroscience of tinnitus: understanding abnormal and normal auditory perception. Front Syst Neurosci. 2012 Jul 11;6:53. doi: 10.3389/fnsys.2012.00053. eCollection 2012. No abstract available. PMID 22798948
- [Background] Atik A. Pathophysiology and treatment of tinnitus: an elusive disease. Indian J Otolaryngol Head Neck Surg. 2014 Jan;66(Suppl 1):1-5. doi: 10.1007/s12070-011-0374-8. Epub 2011 Dec 15. PMID 24533352
- [Background] Sheldrake J, Diehl PU, Schaette R. Audiometric characteristics of hyperacusis patients. Front Neurol. 2015 May 15;6:105. doi: 10.3389/fneur.2015.00105. eCollection 2015. PMID 26029161
- [Background] Sanchez TG, Medeiros IR, Levy CP, Ramalho Jda R, Bento RF. Tinnitus in normally hearing patients: clinical aspects and repercussions. Braz J Otorhinolaryngol. 2005 Jul-Aug;71(4):427-31. doi: 10.1016/s1808-8694(15)31194-0. Epub 2005 Dec 15. PMID 16446955
- [Background] Baguley D, McFerran D, Hall D. Tinnitus. Lancet. 2013 Nov 9;382(9904):1600-7. doi: 10.1016/S0140-6736(13)60142-7. Epub 2013 Jul 2. PMID 23827090